CLINICAL TRIAL: NCT05662904
Title: Genetic Ablation of CD33 in Hematopoietic Stem Cells to Broaden the Therapeutic Index of CD33-directed Immunotherapy in Patients with Acute Myeloid Leukemia (AML)
Brief Title: Genetic Ablation of CD33 in HSC to Broaden the Therapeutic Index of CD33-directed Immunotherapy in Patients with AML
Acronym: GALAXY33
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: University Hospital Heidelberg (Other); University Hospital Dresden (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-002
Record Dates: First submitted 2022-12-06; First posted 2022-12-23 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia (AML)
Keywords: AML; allogeneic stem cell transplantation; gene editing; chemotherapy resistance
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Donor-derived CD33-deleted CD34+ HSC combined with Gemtuzumab-Ozogamicin (GO) (Experimental): Patients will be transplanted with CD33-deleted CD34+ HSC derived from the initially matched family donor. Upon HSC engraftment, patients will be treated with escalating doses of the anti-CD33 antibodydrugconjugate Gemtuzumab-Ozogamicin (GO). A conditioning regimen containing GO (d-14, d-11, d-8), Fludarabine 30 mg/m2 (d-6 to d-3) and Melphalan 140mg/m2 (d-2) is used prior to transplantation.
  Interventions: Biological: Donor-derived CD34+ HSC with CRISPR/Cas9-mediated CD33 deletion; Drug: Gemtuzumab Ozogamicin

INTERVENTIONS:
Biological: Donor-derived CD34+ HSC with CRISPR/Cas9-mediated CD33 deletion — CD33-deleted CD34+ hematopoietic stem cells derived from the initially matched family donor
Drug: Gemtuzumab Ozogamicin — Intrapatient intra-individual dose escalation Level 0: GO day 1 Level 1: GO day 1, day 4 Level 2: GO day 1, day 4, day 7 with repetition after 21 to 28 days up to 84 days.

SUMMARY:
The study "GALAXY33" is an open-label, prospective, nonrandomized, one arm phase I clinical trial in which patients with relapsed AML after allogeneic hematopoietic stem cell transplantation will be transplanted with CD33-deleted CD34+ HSC derived from the initially matched family donor.

DETAILED DESCRIPTION:
CRISPR/Cas9-mediated inactivation of CD33 in hematopoietic stem cells (HSC) may broaden the therapeutic index of CD33-directed immunotherapy for patients with AML by rendering healthy hematopoietic stem and progenitor cells (HSPC) resistant to escalating doses and/or shorter dosing intervals of the CD33-specific antibody-drug conjugate (ADC) Gemtuzumab-ozogamicin (GO).

In this proof of concept trial, we will develop a platform for genome editing of CD34+ HSC and demonstrate the feasibility, safety and efficacy of this approach for targeted therapy of AML.

Upon implementation, the platform shall be used for innovative clinical trials in diverse types of cancer. Outside of leukemias, autologous HSC could be used to ease the procedure.

Patients with relapsed AML after allogeneic hematopoietic stem cell transplantation will be transplanted with CD33-deleted CD34+ HSC derived from the initially matched family donor.

Upon HSC engraftment, patients will be treated with escalating doses of the anti-CD33 antibodydrug conjugate Gemtuzumab-Ozogamicin (GO). A conditioning regimen containing GO (d-14, d-11, d-8),Fludarabine 30 mg/m2 (d-6 to d-3) and Melphalan 140mg/m2 (d-2) is used prior to transplantation.

The clinical trial will be conducted at two trial sites in the University Hospitals in Heidelberg and Dresden.

25 patients will be assessed for eligibility and 12 patients will be allocated into the trial.

ELIGIBILITY:
Key Inclusion Criteria:

* confirmed AML according to the WHO classification
* relapsed disease after allo-SCT from an HLA-identical family donor (≥ 2 months after allo-SCT at time of inclusion)
* ≤ 29% of bone marrow blasts as detected by cytomorphology or immunohistochemistry
* age ≥ 18 years
* confirmed CD33 expression on leukemic blasts at current relapse (as detected by flow cytometry)
* adequate organ function:

  * Renal function defined as: serum creatinine of ≤ 2x ULN or eGFR ≥ 30 mL/min/1.73 m2
  * Liver function defined as:

    * ALT ≤ 3 times the ULN for the respective age
    * Bilirubin ≤ 2.0 mg/dl with the exception of patients with hyperbilirubinemia explained by Gilbert-Meulengracht syndrome (may be included if total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN) or extrahepatic disease (e.g. chronic hemolytic anemia)
* Minimum level of pulmonary reserve defined as ≤ grade 1 dyspnea and pulse oxygenation > 90% on room air
* Hemodynamic stability and LVEF ≥ 40% as confirmed by echocardiogram
* Absolute lymphocyte count (ALC) ≥ 100/mm3

Key Exclusion Criteria:

* ECOG performance status >2
* Confirmed CNS involvement
* Acute or chronic Graft versus Host disease (GvHD)
* Availability of other curative standard treatment options
* Prior treatment with GO
* Prior hepatic veno-occlusive disease (VOD) or sinusoidal obstruction syndrome (SOS)
* Uncontrolled active hepatitis B or C
* HIV-positivity
* Uncontrolled bacterial, viral or fungal infection
* Participation in another clinical trial at the time of screening
* Organ dysfunction (liver, kidney, lung, heart) that is a contraindication for conditioning therapy
* Severe concomitant disease (e.g. uncontrolled arterial hypertension, heart failure NYHA III-IV, uncontrolled diabetes mellitus, uncontrolled hyperlipidemia)
* Unstable angina and/or myocardial infarction within 3 months prior to screening
* Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2028-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
engraftement of gene edited CD34+HSC | on day 28
  successful engraftement of gene edited CD34+HSC in the bone marrow
dose-limiting toxicity | until EOS (day 90)
  dose-limiting toxicity (DLT) of Gemtuzumab-Ozogamicin
toxicities according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0) | until EOS (day 90)
  frequency and grade of AEs with gene-edited HSC transplantation

SECONDARY OUTCOMES:
Anti-tumor efficacy of study treatment in patients with dCD33+ relapsed AML after allo-SCT | until EOS (day 90)
  overall response rate (ORR), complete response (CR), partial response (PR)) at day 90 (EOS) after last GO application)
Time to response | until EOS (day 90)
  Time to response (at least partial response) after the last GO application
Overall response | until EOS (day 90)
  Duration of overall response (DOR) after the last GO application
Progression-free survival | until EOS (day 90)
  Progression-free survival (PFS) after the last GO application
Overall survival | until EOS (day 90)
  Overall survival (OS) after the last GO application
Number of circulating gene edited cells | at screening and days 14, 28, 56, 90
  Number of circulating gene edited cells in the bone marrow and peripheral blood as determined by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Tim Sauer, Dr. med., Principal Investigator — University Hospital Heidelberg
Locations (2):
- Germany (2):
  - University Hospital Dresden, Department of Medicine I, Dresden
  - University Hospital Heidelberg, Internal Medicine V, Heidelberg

IPD SHARING:
Plan to Share IPD: No